CLINICAL TRIAL: NCT04684329
Title: the Value of Serum Esnophilic Cationic Protein as a Diagnostic Parameter in Infants With Cow Milk Protein Allergy
Brief Title: Serum Esnophilic Cationic Protein Level as Diagnostic Marker in Cow Milk Protein Allergy Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed abdelsalam mohamed, doctor, Assiut University
Other Study IDs: cow milk protein allergy
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Characterize the degree of the activation of serum eosinophilc cationic protein (sECP) by measuring its level and establishing whether it is a useful parameter in monitoring oral cow's milk allergy Measure the MPV and NLR levels in infants with CMPA and to determine the suitability of these parameters as biomarkers in diagnosis of CMPA.

DETAILED DESCRIPTION:
Cow's milk protein allergy (CMPA) is the most common cause of food allergies in children with incidence estimated as 2% to 7.5% in the first year of life and is characterized by an inflammatory reaction to milk proteins, Formula and exclusively breast-fed babies can develop CMPA.

The immunologic mechanism behind the development of CMPA is not yet clear. However, it is clear that CMPA is caused by IgE- as well as non-IgE-mediated immune reactions, IgE-mediated CMPA is better described and it is typically immediate, type 1 hypersensitivity (minutes to 2 hours after consumption of cow's milk) while non IgE- mediated CMPA is delayed, type 4 hypersensitivity. a diverse range of symptoms of variable intensity in infants.

Combinations of immediate and delayed reactions to the same allergen may occur in the same patient, symptoms and signs related to CMPA may involve many different organ systems, mostly the skin and the gastro- intestinal and respiratory tracts. The involvement of two systems increases the probability of CMPA, whereas some symptoms are more likely to be present in infant with a positive test for CMP-specific IgE (eg, angioedema, atopic eczema); however, there is a large overlap. The same symptoms may appear in CMP IgE-positive and IgE-negative patients, particularly in infant with gastrointestinal manifestations.

Studies in unselected infants with CMPA show that approximately half of them have atopic eczema, and 25% to 50% are affected by some gastrointestinal tract involvement whereas other clinical manifestations are less common.

It is important to accurately diagnose CMPA to avoid the consequences of either under- or overdiagnosis, skin prick test and serum specific IgE tests are helpful for diagnosis, mainly in IgE-mediated forms . On the other hand, in cases of CMPA with gastrointestinal chronic signs and symptoms, skin prick test and specific IgE tests are usually negative.

This is the reason why the only reliable method of diagnosis in such cases is a food challenge that need to be done in hospital and could be also dangerous, this explain why there is a growing interest to find new biomarkers for diagnosis and follow up.Eosinophil cationic protein (ECP) is a cytotoxic protein released from eosinophils upon activation the measurement of ECP levels can be used as a non invasive indicator to detect active inflammation in the body.

ELIGIBILITY:
Inclusion Criteria:

- All infants (0-12 month) suspected with CMPA

Exclusion Criteria:

* Infants with genetic, metabolic, haematological, or infectious (e.g. :infectious gastroenteritis) diseases will be excluded from the study

Max Age: 12 Months | Sex: All
Age Groups: Child
Study Population: All infants (0-12 month) suspected with CMPA
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, and Overall accuracy value of sECP in CMPA. | one year
  Sensitivity, specificity, and Overall accuracy value of sECP in CMPA.

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university, Asyut, Assuit, Egypt